CLINICAL TRIAL: NCT04596800
Title: Prehabilitation Plus Enhanced Recovery After Surgery Versus Enhanced Recovery After Surgery in Gynecologic Oncology: a Randomized Clinical Trial
Brief Title: Prehabilitation Plus ERAS Versus ERAS in Gynecologic Oncology: a Randomized Clinical Trial
Acronym: PROPER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, André Lopes, MD, Instituto Brasileiro de Controle do Cancer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 36924620.7.0000.0072
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Cancer; Enhanced Recovery After Surgery
Keywords: Prehabilitation; Gynecologic Cancer; ERAS - Enhanced Recovery After Surgery; Gynecologic Surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery; Preoperative Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single-Blind (surgeons and anesthesiologists)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation + Enhanced Recovery After Surgery (Experimental): Patients allocated to the intervention group will undergo prehabilitation protocol (nutrition + exercise + psychological counselling), with individualized monitoring by the multidisciplinary team.
  Interventions: Other: Prehabilitation Program + Enhanced Recovery After Surgery
- Enhanced Recovery After Surgery (Active Comparator): Patients allocated to the control group will not undergo any pre-surgical intervention, except for preoperative counselling, already implicated in ERAS®.
  Interventions: Other: Enhanced Recovery After Surgery

INTERVENTIONS:
Other: Prehabilitation Program + Enhanced Recovery After Surgery — Prehabilitation Program (nutrition + exercise + psychological counseling) + ERAS protocol
  Other Names: Prehabilitation + ERAS
  Arms: Prehabilitation + Enhanced Recovery After Surgery
Other: Enhanced Recovery After Surgery — ERAS
  Other Names: ERAS protocol
  Arms: Enhanced Recovery After Surgery

SUMMARY:
Prospective, interventionist, controlled and randomized study to test the effectiveness of a multimodal prehabilitation protocol in patients who will undergo gynecological surgery.

DETAILED DESCRIPTION:
Prospective, interventionist and randomized controlled trial in a 1: 1 ratio, open to multidisciplinary team and blind to surgeons and anaesthesiologists. The aim is test the effectiveness of a multimodal prehabilitation protocol in patients who will undergo gynecological surgery.

The multidisciplinary prehabilitation program will be applied to the intervention group. For the group participating in the prehabilitation and for the control group, specific recommendations for gynecological cancer defined by the Enhanced Recovery After Surgery (ERAS®) guidelines will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the Informed Consent Form, indicating that they understand the study procedures and their purpose;
* Women aged between 18 and 80 years old;
* Gynecological surgery performed by laparotomy;
* Patients with Eastern Cooperative Oncology Group Performance Status of at least 2 (ECOG ≤2);
* Preoperative schedule that allows prehabilitation intervention for 2 to 3 weeks

Exclusion Criteria:

* Patients under 18 or older than 80 years old;
* ECOG ≥3;
* Significant comorbidities, such as: neurological or musculoskeletal disorder, heart disease and / or respiratory failure that prohibit physical exercise;
* Limitation of ambulation preventing the patient to perform physical exercises;
* Cognitive deterioration or patients with psychiatric disorder that prevents adherence to the program;
* Emergency or urgency surgeries;
* Surgeries by minimally invasive approach (laparoscopy or robotics);
* Vulvectomy or soft tissue surgery without abdominal approach;
* Minor gynaecological surgeries such as conizations;
* Surgeries performed together with other specialties, in which the gynecology team is not primarily responsible for postoperative care;
* If surgery is performed 21 days after the last day of the prehabilitation program, for any reason

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 194 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery time | Up to 30 postoperative days
  Postoperative day patient is ready for discharge, defined as the day the patient has the ability to walk alone, take care of herself, and ingest at least 75% of the daily caloric needs

SECONDARY OUTCOMES:
Complications and Adverse Effects | Up to 30 postoperative days
  Complications and Adverse Effects according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 2017
Readmissions | Up to 30 postoperative days
  Readmission to the Hospital Facilities
Intensive Care Unit admission rates | Up to 30 postoperative days
  Postoperative Intensive Care Unit admission and stay
Health-related Quality of Life | At Baseline, the week before surgery, then at postoperative days 7, 30 and 60
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Compliance to the ERAS® program guideline | Up to 30 postoperative days
  Compliance to ERAS® protocol and implementation of the program
Changes in anxiety and depression from baseline | At Baseline, the week before surgery, then at postoperative days 7, 30 and 60
  Changes in anxiety and depression will be examined using the Hospital Anxiety and Depression Scale. Scores for each sub scale (depression and anxiety) are summed-up and range from 0 to 21. Values from 0-7 indicate normal levels, 8-10 are border values and values from 11-21 are considered to be pathological.
Changes in functional capacity from baseline | At Baseline, the week before surgery, then at postoperative days 30 and 60
  Patients will perform a 6-Minute Walk Test
Change in muscle strength | At Baseline, the week before surgery, then at postoperative days 30 and 60
  Muscle strength is measured by using an dynamometer
Change in body mass | At Baseline, the week before surgery, then at postoperative days 30 and 60
  Body mass is measured by using a bioelectrical impedance analysis
Hospital stay | Up to 30 days
  Days from surgical procedure to hospital discharge
Use of opioids in acute postoperative pain | Up to 30 days
  Use and dosage of opioids in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lopes, MD, Principal Investigator — Instituto Brasileiro de Controle do Cancer
Locations (1):
- Instituto Brasileiro de Controle do Cancer - IBCC, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After publication of the results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study enrollment
Access Criteria: Public

REFERENCES:
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Santa Mina D, Clarke H, Ritvo P, Leung YW, Matthew AG, Katz J, Trachtenberg J, Alibhai SM. Effect of total-body prehabilitation on postoperative outcomes: a systematic review and meta-analysis. Physiotherapy. 2014 Sep;100(3):196-207. doi: 10.1016/j.physio.2013.08.008. Epub 2013 Nov 13. PMID 24439570
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665
- [Background] Iyer R, Gentry-Maharaj A, Nordin A, Burnell M, Liston R, Manchanda R, Das N, Desai R, Gornall R, Beardmore-Gray A, Nevin J, Hillaby K, Leeson S, Linder A, Lopes A, Meechan D, Mould T, Varkey S, Olaitan A, Rufford B, Ryan A, Shanbhag S, Thackeray A, Wood N, Reynolds K, Menon U. Predictors of complications in gynaecological oncological surgery: a prospective multicentre study (UKGOSOC-UK gynaecological oncology surgical outcomes and complications). Br J Cancer. 2015 Feb 3;112(3):475-84. doi: 10.1038/bjc.2014.630. Epub 2014 Dec 23. PMID 25535730
- [Background] Miralpeix E, Mancebo G, Gayete S, Corcoy M, Sole-Sedeno JM. Role and impact of multimodal prehabilitation for gynecologic oncology patients in an Enhanced Recovery After Surgery (ERAS) program. Int J Gynecol Cancer. 2019 Oct;29(8):1235-1243. doi: 10.1136/ijgc-2019-000597. Epub 2019 Aug 30. PMID 31473663
- [Derived] Lopes A, Yamada AMTD, Cardenas TC, Carvalho JN, Oliveira EA, Silva MERD, Andrade JFM, de Souza Neto E, Barros LADR, Costa RLR. PROPER-PRehabilitatiOn Plus Enhanced Recovery after surgery versus enhanced recovery after surgery in gynecologic oncology: a randomized clinical trial. Int J Gynecol Cancer. 2022 Feb;32(2):195-197. doi: 10.1136/ijgc-2021-003170. Epub 2021 Nov 8. PMID 34750197